CLINICAL TRIAL: NCT06067152
Title: REcruitment MAneuvers and Mechanical Ventilation Guided by EIT in Pediatric Acute Respiratory Distress Syndrome (pARDS)
Brief Title: REcruitment MAneuvers and Mechanical Ventilation Guided by EIT in pARDS
Acronym: REMAV-EIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: REMAV-EIT
Record Dates: First submitted 2022-09-08; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-08

CONDITIONS: ARDS; Pediatric Respiratory Distress Syndrome; Respiratory Disease
Keywords: Non invasive ventilation; electrical impedance tomography;
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiration Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T0= Enrollment (Active Comparator): mechanical ventilation will be set according to the standard of care criteria
  Interventions: Device: EIT measurement
- T1= guided MV at the end of SRM trial (Active Comparator): EIT guided mechanical ventilation will be set
  Interventions: Device: Staircase Recruitment Maneuvers with EIT guided and decremental PEEP trial; Device: Setting of EIT-guided mechanical ventilation
- T2= 24 hours with EIT guided MV (Active Comparator): evaluation of mechanical ventilation after 24h EIT-guided ventilation
  Interventions: Device: Reevaluation after 24 h

INTERVENTIONS:
Device: EIT measurement — Evaluation of mechanical ventilation and ventilation distribution through EIT. Mechanical ventilation is set by the physician according to clinical protocolized criteria
  Arms: T0= Enrollment
Device: Staircase Recruitment Maneuvers with EIT guided and decremental PEEP trial — SRMs will be performed with a standardized ventilation protocol. Patient will be sedated, paralyzed and ventilated in pressure controlled mode, FIO2 to obtain SPO2> 92%, RR 25, I:E =1:1.5. Alarm of pressure limit will be set at 35 cmH2O. The ventilator will be equipped with inspiratory and expiratory hold taste. Inspiratory and expiratory occlusion will be held for 5 seconds, data will be stored and analyzed with the ventilator own tool.
  Decremental PEEP trial will start if plateau pressure 30 cmH2O will be reached or end inspiratory transpulmonary pressure will exceed 28 cmH2O value. Once reached this level of plateau or transpulmonary pressure, PEEP will be reduced in three steps from 12, 10 and finally to 8 cmH2O every 20 minutes
  Other Names: SRMs EIT-guided and DP trial
  Arms: T1= guided MV at the end of SRM trial
Device: Setting of EIT-guided mechanical ventilation — Mechanical ventilation is set according to EIT measurement
  Arms: T1= guided MV at the end of SRM trial
Device: Reevaluation after 24 h — Evaluation of mechanical ventilation and ventilation distribution through EIT after 24h of ventilation EIT-guided
  Arms: T2= 24 hours with EIT guided MV

SUMMARY:
There is evidence from randomized controlled trials in adult patients with Acute Respiratory Distress Syndrome (ARDS) suggesting that delivering small tidal volumes with adequate levels of Positive End-Expiratory Pressure (PEEP) and a restrictive fluid strategy could improve outcome. However, there are data and common bedside experience that individual patients may or may not respond to interventions, such as escalation of PEEP or positional changes, and there may be a role for a more personalized ventilator strategy.

This strategy could account for the unique individual morphology of lung disease, such as the amount of atelectasis and overdistension as a percentage of total lung tissue, the exact location of atelectasis, and whether positional changes or elevation of PEEP produce lung recruitment or overdistension.

Stepwise Recruitment maneuvers (SRMs) in pARDS improve oxygenation in majority of patients. SRMs should be considered for use on an individualized basis in patients with pARDS should be considered if SpO2 decreases by ≥ 5% within 5 minutes of disconnection during suction or coughing or agitation. If a recruitment maneuver is conducted, a decremental PEEP trial must be done to determine the minimum PEEP that sustains the benefits of the recruitment maneuver.

Electrical impedance tomography (EIT), a bedside monitor to describe regional lung volume changes, displays a real-time cross-sectional image of the lung. EIT is a non-invasive, non-operator dependent, bedside, radiations-free diagnostic tool, feasible in paediatric patients and repeatable. It allows to study ventilation distribution dividing lungs in four Region Of Interest (ROI), that are layers distributed in an anteroposterior direction, and shows how ventilation is distributed in the areas concerned.

EIT measures and calculates other parameters that are related not only to the distribution of ventilation, but also to the homogeneity of ventilation and the response to certain therapeutic maneuvers, such as SRMs or PEEP-application.

Aim of this study is to provide a protocolized strategy to assess optimal recruitment and PEEP setting, tailored on the patients individual response in pARDS.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and mechanically ventilated children, ageing 1 months-5 years and meeting the PALICC definition for pediatric Acute Respiratory Distress Syndrome (pARDS)
* Informed Consent signed

Exclusion Criteria: Patients with one or more of the following characteristics:

* Previous barotrauma (pneumothorax, pneumomediastinum or subcutaneous emphysema)
* Signs of intracranial hypertension
* Cyanotic congenital cardiac disease
* Dorso-lumbar pathologies or other bone pathologies associated with restrictive lung disease (such as scoliosis, kyphosis)
* Implantable devices not compatible with EIT (such as pace-makers and implantable cardioverter defibrillator)
* Controindication to positioning the esophageal catheter (surgery, esophageal stenosis)

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Regional Ventilation Delay, RDV (pixels %), at T2 and T0 | 1 day
  RDV is an index of atelectrauma, supra-distention and in general an inhomogeneous ventilation

SECONDARY OUTCOMES:
Differences in Tidal Impedance Distribution,TID (pixels %), at T0, T1 and T2 | 1 day
  for every breathing cycle, a so-called tidal image is generated and each pixel of represents the difference in impedance between end-inspiration and end-expiration. The median value of each tidal image is calculated for the lung area
Gravity Centre, GC, differences (pixels %) at T0, T1 and T2 | 1 day
  it is the weighted mean of row sums obtained from TV image and it indicates ventral-to-dorsal shifts in ventilation distribution due to lung opening and closing
Respiratory Rate at T0, T1 and T2 | 1 day
  Respiratory rate (breaths/min)
FiO2 (%) at T0, T1 and T2 | 1 day
  FiO2 (%)
Respiratory compliance at T0, T1 and T2 | 1 day
  Respiratory System Compliance
Lung compliance at T0, T1 and T2 | 1 day
  Clung Lung compliance
Chest Wall compliance at T0, T1 and T2 | 1 day
  Chest Wall compliance
S/F ratio at T0, T1 and T2 | 1 day
  S/F ratio
Sistolic Blood Pressure at T0, T1 and T2 | 1 day
  SBP (mmHg)
Diastolic Blood Pressure at T0, T1 and T2 | 1 day
  DBP (mmHg)
pH at T0, T1 and T2 | 1 day
  pH
SpO2 at T0, T1 and T2 | 1 day
  SpO2 (%)
PaO2 at T0, T1 and T2 | 1 day
  PaO2 (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Chidini, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Result] Briel M, Meade M, Mercat A, Brower RG, Talmor D, Walter SD, Slutsky AS, Pullenayegum E, Zhou Q, Cook D, Brochard L, Richard JC, Lamontagne F, Bhatnagar N, Stewart TE, Guyatt G. Higher vs lower positive end-expiratory pressure in patients with acute lung injury and acute respiratory distress syndrome: systematic review and meta-analysis. JAMA. 2010 Mar 3;303(9):865-73. doi: 10.1001/jama.2010.218. PMID 20197533
- [Result] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- [Result] Wolf GK, Gomez-Laberge C, Kheir JN, Zurakowski D, Walsh BK, Adler A, Arnold JH. Reversal of dependent lung collapse predicts response to lung recruitment in children with early acute lung injury. Pediatr Crit Care Med. 2012 Sep;13(5):509-15. doi: 10.1097/PCC.0b013e318245579c. PMID 22622650
- [Result] Gattinoni L, Caironi P, Cressoni M, Chiumello D, Ranieri VM, Quintel M, Russo S, Patroniti N, Cornejo R, Bugedo G. Lung recruitment in patients with the acute respiratory distress syndrome. N Engl J Med. 2006 Apr 27;354(17):1775-86. doi: 10.1056/NEJMoa052052. PMID 16641394
- [Result] Papazian L, Forel JM, Gacouin A, Penot-Ragon C, Perrin G, Loundou A, Jaber S, Arnal JM, Perez D, Seghboyan JM, Constantin JM, Courant P, Lefrant JY, Guerin C, Prat G, Morange S, Roch A; ACURASYS Study Investigators. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010 Sep 16;363(12):1107-16. doi: 10.1056/NEJMoa1005372. PMID 20843245
- [Result] Gattinoni L, Tognoni G, Pesenti A, Taccone P, Mascheroni D, Labarta V, Malacrida R, Di Giulio P, Fumagalli R, Pelosi P, Brazzi L, Latini R; Prone-Supine Study Group. Effect of prone positioning on the survival of patients with acute respiratory failure. N Engl J Med. 2001 Aug 23;345(8):568-73. doi: 10.1056/NEJMoa010043. PMID 11529210
- [Result] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Result] Victorino JA, Borges JB, Okamoto VN, Matos GF, Tucci MR, Caramez MP, Tanaka H, Sipmann FS, Santos DC, Barbas CS, Carvalho CR, Amato MB. Imbalances in regional lung ventilation: a validation study on electrical impedance tomography. Am J Respir Crit Care Med. 2004 Apr 1;169(7):791-800. doi: 10.1164/rccm.200301-133OC. Epub 2003 Dec 23. PMID 14693669
- [Result] Wrigge H, Zinserling J, Muders T, Varelmann D, Gunther U, von der Groeben C, Magnusson A, Hedenstierna G, Putensen C. Electrical impedance tomography compared with thoracic computed tomography during a slow inflation maneuver in experimental models of lung injury. Crit Care Med. 2008 Mar;36(3):903-9. doi: 10.1097/CCM.0B013E3181652EDD. PMID 18431279
- [Result] Wolf GK, Gomez-Laberge C, Rettig JS, Vargas SO, Smallwood CD, Prabhu SP, Vitali SH, Zurakowski D, Arnold JH. Mechanical ventilation guided by electrical impedance tomography in experimental acute lung injury. Crit Care Med. 2013 May;41(5):1296-304. doi: 10.1097/CCM.0b013e3182771516. PMID 23474677
- [Result] Zhao Z, Moller K, Steinmann D, Frerichs I, Guttmann J. Evaluation of an electrical impedance tomography-based Global Inhomogeneity Index for pulmonary ventilation distribution. Intensive Care Med. 2009 Nov;35(11):1900-6. doi: 10.1007/s00134-009-1589-y. Epub 2009 Aug 4. PMID 19652949
- [Result] Spinelli E, Mauri T, Fogagnolo A, Scaramuzzo G, Rundo A, Grieco DL, Grasselli G, Volta CA, Spadaro S. Correction to: Electrical impedance tomography in perioperative medicine: careful respiratory monitoring for tailored interventions. BMC Anesthesiol. 2019 Sep 4;19(1):172. doi: 10.1186/s12871-019-0840-5. PMID 31481006
- [Result] Pediatric Acute Lung Injury Consensus Conference Group. Pediatric acute respiratory distress syndrome: consensus recommendations from the Pediatric Acute Lung Injury Consensus Conference. Pediatr Crit Care Med. 2015 Jun;16(5):428-39. doi: 10.1097/PCC.0000000000000350. PMID 25647235
- [Result] Kneyber MCJ, de Luca D, Calderini E, Jarreau PH, Javouhey E, Lopez-Herce J, Hammer J, Macrae D, Markhorst DG, Medina A, Pons-Odena M, Racca F, Wolf G, Biban P, Brierley J, Rimensberger PC; section Respiratory Failure of the European Society for Paediatric and Neonatal Intensive Care. Recommendations for mechanical ventilation of critically ill children from the Paediatric Mechanical Ventilation Consensus Conference (PEMVECC). Intensive Care Med. 2017 Dec;43(12):1764-1780. doi: 10.1007/s00134-017-4920-z. Epub 2017 Sep 22. PMID 28936698
- [Result] Chiumello D, Carlesso E, Cadringher P, Caironi P, Valenza F, Polli F, Tallarini F, Cozzi P, Cressoni M, Colombo A, Marini JJ, Gattinoni L. Lung stress and strain during mechanical ventilation for acute respiratory distress syndrome. Am J Respir Crit Care Med. 2008 Aug 15;178(4):346-55. doi: 10.1164/rccm.200710-1589OC. Epub 2008 May 1. PMID 18451319
- [Result] Protti A, Cressoni M, Santini A, Langer T, Mietto C, Febres D, Chierichetti M, Coppola S, Conte G, Gatti S, Leopardi O, Masson S, Lombardi L, Lazzerini M, Rampoldi E, Cadringher P, Gattinoni L. Lung stress and strain during mechanical ventilation: any safe threshold? Am J Respir Crit Care Med. 2011 May 15;183(10):1354-62. doi: 10.1164/rccm.201010-1757OC. Epub 2011 Feb 4. PMID 21297069
- [Result] Chiumello D, Cressoni M, Colombo A, Babini G, Brioni M, Crimella F, Lundin S, Stenqvist O, Gattinoni L. The assessment of transpulmonary pressure in mechanically ventilated ARDS patients. Intensive Care Med. 2014 Nov;40(11):1670-8. doi: 10.1007/s00134-014-3415-4. Epub 2014 Aug 12. PMID 25112501
- [Result] Turner DA, Heitz D, Zurakowski D, Arnold JH. Automated measurement of the lower inflection point in a pediatric lung model. Pediatr Crit Care Med. 2009 Jul;10(4):511-6. doi: 10.1097/PCC.0b013e3181a0e274. PMID 19325511
- [Result] Rosemeier I, Reiter K, Obermeier V, Wolf GK. Mechanical Ventilation Guided by Electrical Impedance Tomography in Children With Acute Lung Injury. Crit Care Explor. 2019 Jul 1;1(7):e0020. doi: 10.1097/CCE.0000000000000020. eCollection 2019 Jul. PMID 32166264
- [Result] Cruces P, Donoso A, Valenzuela J, Diaz F. Respiratory and hemodynamic effects of a stepwise lung recruitment maneuver in pediatric ARDS: a feasibility study. Pediatr Pulmonol. 2013 Nov;48(11):1135-43. doi: 10.1002/ppul.22729. Epub 2012 Dec 19. PMID 23255291
- [Result] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Result] Stapleton RD, Suratt BT, Neff MJ, Wurfel MM, Ware LB, Ruzinski JT, Caldwell E, Hallstrand TS, Parsons PE. Bronchoalveolar fluid and plasma inflammatory biomarkers in contemporary ARDS patients. Biomarkers. 2019 Jun;24(4):352-359. doi: 10.1080/1354750X.2019.1581840. Epub 2019 Mar 4. PMID 30744430
- See also: National Heart, Lung, and Blood Institute ARDS Clinical Trials Network: Mechanical Ventilation Protocol Summary. 2008 — http://www.ardsnet.org/files/ventilator_protocol_2008-07.pdf